CLINICAL TRIAL: NCT00784134
Title: Clot Lysis: Evaluating Accelerated Resolution of Intraventricular Hemorrhage Phase III
Acronym: CLEAR III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Genentech, Inc. (Industry); Emissary International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVH06; 5U01NS062851-05 (NIH)
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Intraventricular Hemorrhage
Keywords: intraventricular hemorrhage thrombolysis
MeSH Terms: interventions — Tissue Plasminogen Activator; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alteplase (Experimental): administration of alteplase via the intraventricular catheter
  Interventions: Drug: Alteplase
- Saline Placebo (Placebo Comparator): 1 ml of normal saline administered via the intraventricular catheter
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Alteplase — 1.0 mg of alteplase will be administered via the intraventricular catheter every 8 hours for up to 12 doses
  Other Names: Cathflo Activase; rt-PA
  Arms: Alteplase
Other: Normal saline — 1 ml of normal saline will be administered via the intraventricular catheter every 8 hours for up to 12 doses
  Arms: Saline Placebo

SUMMARY:
The overall objective of this Phase III clinical trial is to obtain information from a population of 500 ICH subjects with intraventricular hemorrhage (IVH), representative of current clinical practice and national demographics of ICH regarding the benefit (or lack thereof) of IVH clot removal on subject function as measured by modified Rankin Scale (mRS). This application requests funding for five years to initiate a Phase III randomized clinical trial (RCT) testing the benefit of clot removal for intraventricular hemorrhage. The investigators propose to compare extraventricular drainage (EVD) use plus recombinant tissue plasminogen activator (rt-PA; Alteplase; Genentech, Inc., San Francisco, CA) with EVD+ placebo in the management and treatment of subjects with small intracerebral hemorrhage (ICH) and large intraventricular hemorrhage (IVH defined as ICH < 30 cc and obstruction of the 3rd or 4th ventricles by intraventricular blood clot).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Symptom onset less than 24 hrs prior to diagnostic CT scan
* Spontaneous ICH less than or equal to 30 cc or primary IVH
* IVH obstructing 3rd and/or 4th ventricles
* ICH clot stability at 6 hours or more post IVC placement
* IVH clot stability at 6 hours or more post IVC placement
* Catheter tract bleeding stability 6 hours or more post IVC placement
* EVD placed per standard medical care
* SBP less than 200 mmHg sustained for 6 hours prior to drug administration
* Able to randomize within 72 hours of diagnostic CT scan
* Historical Rankin of 0 or 1

Exclusion Criteria:

* Suspected or untreated ruptured cerebral aneurysm, AVM, or tumor
* Presence of a choroid plexus vascular malformation or Moyamoya
* Clotting disorders
* Platelet count less than 100,000, INR greater than 1.4
* Pregnancy
* Infratentorial hemorrhage
* SAH at clinical presentation
* ICH/IVH enlargement that cannot be stabilized in the treatment time window
* Ongoing internal bleeding
* Superficial or surface bleeding
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Planned or simultaneous participation (between screening and Day-30) in another interventional medical investigation or clinical trial.
* No subject or legal representative to give written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2009-07; Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F. Hanley, MD, Study Chair — Johns Hopkins University
Locations (81):
- United States (52):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Arizona, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Southern California - Keck School of Medicine, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Intercoastal Medical Center, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Rush University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Ruan Neurology Clinical and Research Center, Des Moines, Iowa
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - St. Luke's Brain and Stroke Institute, Kansas City, Missouri
  - Springfield Neurological and Spine Institute, Springfield, Missouri
  - St. Louis University, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - New Jersey Neuroscience Institute at JFK, Edison, New Jersey
  - University of Buffalo, Buffalo, New York
  - Northshore University Hospital Long Island, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University, New York, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case-Western Reserve University Hospital, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Maine Medical Center, Portland, Oregon
  - Providence Stroke Center, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt, Nashville, Tennessee
  - University of Texas, Southwestern, Dallas, Dallas, Texas
  - University of Texas, Houston, Houston, Texas
  - University of Texas, San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Brazil (5):
  - Hospital Sao Jose, Joinville, Joinville, Santa Catarina
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital de Pronto Socorro de Porto Alegre, Porto Alegre
  - Hospital de Clinicas de Ribeirao Preto, Ribeirão Preto
  - Hospital Sao Paulo Universidade Federal de Sao Paulo / UNIFESP, São Paulo
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Montreal Neurological Institute at McGill University, Montreal, Quebec
- Germany (6):
  - University of Erlangen, Erlangen
  - University of Halle, Halle
  - University of Heidelberg, Heidelberg
  - University of Leipzig, Leipzig
  - University of Mainz, Mainz
  - University of Tubingen, Tübingen
- Hungary (4):
  - University of Szeged, Szeged, Csongrád megye
  - Honved Korhaz, Budapest
  - University of Debrecen, Debrecen
  - University of Pecs, Pécs
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Hebrew University Hospital, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Spain (3):
  - Bellvitge Hospital, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
- Switzerland (2):
  - University of Zurich, Zurich, Canton of Zurich
  - University Hospital, Inselpital, Bern, Bern
- United Kingdom (3):
  - Salford Royal NHS Foundation Trust, Salford, Manchester
  - Newcastle General Hospital, Newcastle upon Tyne
  - University of Southampton Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roh DJ, Asonye IS, Carvalho Poyraz F, Magid-Bernstein JR, Joiner EF, Avadhani R, Awad I, Hanley DF, Ziai WC, Murthy SB. Intraventricular Hemorrhage Expansion in the CLEAR III Trial: A Post Hoc Exploratory Analysis. Stroke. 2022 Jun;53(6):1847-1853. doi: 10.1161/STROKEAHA.121.037438. Epub 2022 Jan 28. PMID 35086362
- [Derived] Hansen BM, Ullman N, Muschelli J, Norrving B, Dlugash R, Avadhani R, Awad I, Zuccarello M, Ziai WC, Hanley DF, Thompson RE, Lindgren A; MISTIE and CLEAR Investigators. Relationship of White Matter Lesions with Intracerebral Hemorrhage Expansion and Functional Outcome: MISTIE II and CLEAR III. Neurocrit Care. 2020 Oct;33(2):516-524. doi: 10.1007/s12028-020-00916-4. PMID 32026447
- [Derived] Porter AL, Ebot J, Lane K, Mooney LH, Lannen AM, Richie EM, Dlugash R, Mayo S, Brott TG, Ziai W, Freeman WD, Hanley DF. Enhancing the Informed Consent Process Using Shared Decision Making and Consent Refusal Data from the CLEAR III Trial. Neurocrit Care. 2020 Feb;32(1):340-347. doi: 10.1007/s12028-019-00860-y. PMID 31571176
- [Derived] Eslami V, Tahsili-Fahadan P, Rivera-Lara L, Gandhi D, Ali H, Parry-Jones A, Nelson LS, Thompson RE, Nekoobakht-Tak S, Dlugash R, McBee N, Awad I, Hanley DF, Ziai WC. Influence of Intracerebral Hemorrhage Location on Outcomes in Patients With Severe Intraventricular Hemorrhage. Stroke. 2019 Jul;50(7):1688-1695. doi: 10.1161/STROKEAHA.118.024187. Epub 2019 Jun 10. PMID 31177984
- [Derived] Fam MD, Zeineddine HA, Eliyas JK, Stadnik A, Jesselson M, McBee N, Lane K, Cao Y, Wu M, Zhang L, Thompson RE, John S, Ziai W, Hanley DF, Awad IA; CLEAR III Trial Investigators. CSF inflammatory response after intraventricular hemorrhage. Neurology. 2017 Oct 10;89(15):1553-1560. doi: 10.1212/WNL.0000000000004493. Epub 2017 Sep 8. PMID 28887375
- [Derived] Hanley DF, Lane K, McBee N, Ziai W, Tuhrim S, Lees KR, Dawson J, Gandhi D, Ullman N, Mould WA, Mayo SW, Mendelow AD, Gregson B, Butcher K, Vespa P, Wright DW, Kase CS, Carhuapoma JR, Keyl PM, Diener-West M, Muschelli J, Betz JF, Thompson CB, Sugar EA, Yenokyan G, Janis S, John S, Harnof S, Lopez GA, Aldrich EF, Harrigan MR, Ansari S, Jallo J, Caron JL, LeDoux D, Adeoye O, Zuccarello M, Adams HP Jr, Rosenblum M, Thompson RE, Awad IA; CLEAR III Investigators. Thrombolytic removal of intraventricular haemorrhage in treatment of severe stroke: results of the randomised, multicentre, multiregion, placebo-controlled CLEAR III trial. Lancet. 2017 Feb 11;389(10069):603-611. doi: 10.1016/S0140-6736(16)32410-2. Epub 2017 Jan 10. PMID 28081952
- [Derived] Webb AJ, Ullman NL, Morgan TC, Muschelli J, Kornbluth J, Awad IA, Mayo S, Rosenblum M, Ziai W, Zuccarrello M, Aldrich F, John S, Harnof S, Lopez G, Broaddus WC, Wijman C, Vespa P, Bullock R, Haines SJ, Cruz-Flores S, Tuhrim S, Hill MD, Narayan R, Hanley DF; MISTIE and CLEAR Investigators. Accuracy of the ABC/2 Score for Intracerebral Hemorrhage: Systematic Review and Analysis of MISTIE, CLEAR-IVH, and CLEAR III. Stroke. 2015 Sep;46(9):2470-6. doi: 10.1161/STROKEAHA.114.007343. Epub 2015 Aug 4. PMID 26243227
- See also: Related Info — http://braininjuryoutcomes.com
- Available data/document: Data repository-VISTA: Data repository-VISTA — http://vista.gla.ac.uk — when available
- Available data/document: Study Protocol — http://vista.gla.ac.uk — when available
- Available data/document: Statistical Analysis Plan — http://vista.gla.ac.uk — when available

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alteplase | Saline Placebo
Started | 249 | 251
Completed | 246 | 245
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alteplase | Saline Placebo | Total
Number analyzed (Participants) | 249 | 251 | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 182 | 172 | 354
  >=65 years | 67 | 79 | 146
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 117 | 222
  Male | 144 | 134 | 278
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 92 | 78 | 170
  White | 144 | 161 | 305
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 6 | 9
  Hungary | 7 | 6 | 13
  United States | 190 | 180 | 370
  Brazil | 1 | 3 | 4
  United Kingdom | 4 | 4 | 8
  Israel | 13 | 24 | 37
  Switzerland | 1 | 3 | 4
  Germany | 21 | 18 | 39
  Spain | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Participants With Modified Rankin Scale (mRS) <=3 - Dichotomized Analysis
Description: Analysis modified on September 29, 2015 to account for adaptive randomization. The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from 0 (perfect health without symptoms) to 6 (death).
Time Frame: 180 days
Population: All the non-missing mRS scores at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 246 | 245
percentage of participants | 47.6 | 44.9
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.554, Chi-squared; Risk Difference (RD) = 0.027, 95% CI 2-sided [-0.062 to 0.115]
Statistical Analysis 2: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.465, Multivariable Logit Model — Multivariable logit model adjusted for age, GCS, thalamus, stability ICH volume and stability IVH volume; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.75 to 1.87]

2. Primary Outcome: Participant Score on the Modified Rankin Scale (mRS) - Ordinal Analysis
Description: The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from 0 (perfect health without symptoms) to 6 (death).
Time Frame: 180 days
Population: All the non-missing mRS scores at 180 days were analyzed.
Measure: Median (Inter-Quartile Range); unit: mRS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 246 | 245
mRS score | 4 [3 to 5] | 4 [3 to 6]
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.484, Generalized ordered Logit Model — Generalized ordered logit model adjusted for age, GCS, thalamus, stability ICH volume and stability IVH volume (categorical) compares odds ratio for mRS score > K v. <= K for K = 1 - 4; Alt v. Sal; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.63 to 1.25]
Statistical Analysis 2: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p < 0.001, Generalized ordered Logit Model — The same generalized ordered logit model, adjusting for age, GCS, thalamus, stability ICH volume and stability IVH volume (categorical), compares odds ratio for mRS score greater than 5 versus mRS score equal or less than 5 (dead versus alive); Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.28 to 0.71]

3. Primary Outcome: Participants With Modified Rankin Scale (mRS) <=4 - Dichotomized Analysis
Description: as for outcome 2
Time Frame: 180 days
Population: All the non-missing mRS scores at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 246 | 245
percentage of participants | 64.2 | 61.6
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.552, Chi-squared; Risk Difference (RD) = 0.026, 95% CI 2-sided [-0.059 to 0.111]
Statistical Analysis 2: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.350, Multivariable Logit Model — Multivariable logit model adjusting for age, GCS, thalamus, stability ICH volume and stability IVH volume (categorical); Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.80 to 1.90]

4. Primary Outcome: Random Effects Assessment of Site Effect on Modified Rankin Scale (mRS) <= 3
Description: as for outcome 2
Time Frame: 180 days
Population: All the non-missing mRS scores at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 246 | 245
percentage of participants | 47.6 | 44.9
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.428, Random Effects Model — Random effects model with site as random effect adjusted for age, GCS, thalamus, stability ICH volume and stability IVH volume (categorical); Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.78 to 1.80]

5. Primary Outcome: Longitudinal Assessment of Participants With Modified Rankin Scale (mRS) <=3
Description: Comparing longitudinal modified Rankin Scale (mRS) scores 0-3 at Day 30 and Day 180. The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from 0 (perfect health without symptoms) to 6 (death).
Time Frame: 30 days and 180 days
Population: All the non-missing mRS scores at 30 days and 180 days were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 246 | 249
Percentage of participants
  Day 30: number analyzed (Participants) | 245 | 249
  Day 30 | 20.4 | 16.5
  Day 180: number analyzed (Participants) | 246 | 245
  Day 180 | 48.0 | 45.7
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Logit mRS scores 0-3 at 30 days; Test type: Superiority or Other; p = 0.384, Generalized Estimating Equation Model; Generalized estimating equation model adjusting for age, GCS, thalamus, stability ICH volume and stability IVH volume (categorical); Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.75 to 2.10]
Statistical Analysis 2: Comparison: Alteplase vs Saline Placebo; Logit mRS scores 0-3 at 180 days; Test type: Superiority or Other; p = 0.964, Generalized Estimating Equation Model; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.62 to 1.64]

6. Secondary Outcome: All Cause Mortality
Time Frame: 180 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
percentage of participants | 18.5 | 29.1
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.0056, Log Rank

7. Secondary Outcome: Clot Removal (Amount of Residual Blood)
Description: Change in blood volume measured between stability scan and end of treatment scan
Time Frame: 72 hours
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: odds ratio per time-weighted ml
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
odds ratio per time-weighted ml | 0.96 | 0.97
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p < 0.001, AUC/ Logit Model

8. Secondary Outcome: Intensity of Critical Care Management - Hospital Days
Description: Intensity of critical care management as measured by hospital and ICU length of stay, frequency of ICP >20 mmHg events, use of mechanical ventilation, pressors, and ventriculoperitioneal shunts, frequency of systemic infections.
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Median (Inter-Quartile Range); unit: Number of days
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
Number of days | 23 [17 to 31] | 24 [16 to 31]
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.771, Kruskal-Wallis

9. Secondary Outcome: Intensity of Critical Care Management - ICU Days
Description: as for outcome 8
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Median (Inter-Quartile Range); unit: Number of days
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
Number of days | 14 [11 to 21] | 15 [12 to 22]
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.098, Kruskal-Wallis

10. Secondary Outcome: Intensity of Critical Care Management - ICP Management
Description: as for outcome 8
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: Percentage of events of ICP >20mmHg
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
Percentage of events of ICP >20mmHg | 9.8 | 10.2
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.450, Generalized Linear Models

11. Secondary Outcome: Intensity of Critical Care Management - Mechanical Ventilation
Description: as for outcome 8
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: % of participants with ventilation
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
% of participants with ventilation | 73.9 | 76.5
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.501, Chi-squared

12. Secondary Outcome: Intensity of Critical Care Management - Pressors
Description: as for outcome 8
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: % of participants with pressors
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
% of participants with pressors | 24.1 | 25.1
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.795, Chi-squared

13. Secondary Outcome: Intensity of Critical Care Management - Shunts
Description: as for outcome 8
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: % of participants with shunts
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
% of participants with shunts | 18.5 | 17.5
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.784, Chi-squared

14. Secondary Outcome: Intensity of Critical Care Management - All Infections
Description: as for outcome 8
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: % of participants with infections
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
% of participants with infections | 48.2 | 50.6
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.592, Chi-squared

15. Secondary Outcome: Intensity of Critical Care Management - Pneumonia
Description: as for outcome 8
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: % of participants with pneumonia
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
% of participants with pneumonia | 26.1 | 32.7
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.105, Chi-squared

16. Secondary Outcome: Intensity of Critical Care Management - All Infections
Description: as for outcome 8
Time Frame: 180 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: % of participants with infections
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
% of participants with infections | 49.8 | 56.2
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.152, Chi-squared

17. Secondary Outcome: Safety/Mortality - Mortality Within 30 Days
Description: Frequency of bacterial brain infections, symptomatic brain bleeds, and mortality.
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: Percentage of patients
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
Percentage of patients | 8.8 | 14.3
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.055, Fisher Exact; Risk Difference (RD) = -0.055, 95% CI 2-sided [-0.111 to 0.008]

18. Secondary Outcome: Safety/Mortality - Bacterial Brain Infections Within 30 Days
Description: Frequency of bacterial brain infections, symptomatic brain bleeds, and mortality.
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: % of participants with brain infection
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
% of participants with brain infection | 6.8 | 10.4
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.202, Fisher Exact; Risk Difference (RD) = -0.035, 95% CI 2-sided [-0.084 to 0.014]

19. Secondary Outcome: Safety/Mortality - Systematic Bleeds Within 72 Hours
Description: Frequency of bacterial brain infections, symptomatic brain bleeds, and mortality.
Time Frame: 72 hours
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: % of participants with systematic bleeds
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
% of participants with systematic bleeds | 2.4 | 2.0
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.771, Fisher Exact; Risk Difference (RD) = 0.004, 95% CI 2-sided [-0.022 to 0.030]

20. Secondary Outcome: Safety/Mortality - Systematic Bleeds Within 30 Days
Description: Frequency of bacterial brain infections, symptomatic brain bleeds, and mortality.
Time Frame: 30 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: % of participants with systematic bleeds
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
% of participants with systematic bleeds | 3.6 | 3.2
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.811, Fisher Exact; Risk Difference (RD) = 0.004, 95% CI 2-sided [-0.028 to 0.036]

21. Secondary Outcome: Adverse and Serious Adverse Events
Description: Assessment of number of adverse and serious adverse events by treatment group.
Time Frame: 180 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
percentage of participants | 45.8 | 60.2
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.0017, Fisher Exact; Risk Difference (RD) = -0.144, 95% CI 2-sided [-0.230 to -0.057]

22. Secondary Outcome: Predicting Hazards of Death by Treatment Group
Description: Cox Proportional Hazards Model is used to predict the hazards ratio by treatment group.
Time Frame: 180 days
Population: All patients that were enrolled in CLEAR III were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 249 | 251
percentage of participants | 18.5 | 29.1
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.006, Cox Proportional Hazards Model; Adjusted Cox Proportional Hazards Model adjusting for age, GCS, thalamus, stability ICH volume and stability IVH volume (categorical); Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.41 to 0.86]

23. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by Race (African-American)
Description: Assessment of modified Rankin Scale (mRS) score 0-3 compared by race, gender, age, IVH size, and ICH location. The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It is scored from 0 (perfect health without symptoms) to 6 (death).
Time Frame: 180 days
Population: All patients that reported they were African-American with a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 90 | 75
Percentage of participants | 54.4 | 48.0
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.410, Chi-squared; Risk Difference (RD) = 0.064, 95% CI 2-sided [-0.088 to 0.217]

24. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by Race (White)
Description: as for outcome 23
Time Frame: 180 days
Population: All patients that reported they were White with a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 143 | 158
percentage of participants | 43.4 | 41.8
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.781, Chi-squared; Risk Difference (RD) = 0.016, 95% CI 2-sided [-0.096 to 0.128]

25. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by Gender (Female)
Description: as for outcome 23
Time Frame: 180 days
Population: All female patients with a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 103 | 114
percentage of participants | 47.6 | 45.6
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.773, Chi-squared; Risk Difference (RD) = 0.020, 95% CI 2-sided [-0.113 to 0.152]

26. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by Gender (Male)
Description: as for outcome 23
Time Frame: 180 days
Population: All male patients with a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 143 | 131
percentage of participants | 47.6 | 44.3
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.587, Chi-squared; Risk Difference (RD) = 0.032, 95% CI 2-sided [-0.085 to 0.151]

27. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by Age (65 Years or Under)
Description: as for outcome 23
Time Frame: 180 days
Population: All patients 65 years of age or under with a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 179 | 167
Percentage of participants | 53.6 | 52.1
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.775, Chi-squared; Risk Difference (RD) = 0.015, 95% CI 2-sided [-0.09 to 0.121]

28. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by Age (Over 65 Years)
Description: as for outcome 23
Time Frame: 180 days
Population: All patients over 65 years of age with a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 67 | 78
Percentage of participants | 31.3 | 29.5
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.808, Chi-squared; Risk Difference (RD) = 0.019, 95% CI 2-sided [-0.132 to 0.169]

29. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by IVH Size (Less Than 20ml)
Description: as for outcome 23
Time Frame: 180 days
Population: All patients with an IVH size less than 20ml and a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 109 | 108
percentage of participants | 55.1 | 58.3
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.625, Chi-squared; Risk Difference (RD) = 0.033, 95% CI 2-sided [-0.165 to 0.099]

30. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by IVH Size (20-50ml)
Description: as for outcome 23
Time Frame: 180 days
Population: All patients with an IVH size between 20ml and 50ml and a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 110 | 109
percentage of participants | 47.3 | 38.5
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.191, Chi-squared; Risk Difference (RD) = 0.087, 95% CI 2-sided [-0.043 to 0.218]

31. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by IVH Size (Greater Than 50ml)
Description: as for outcome 23
Time Frame: 180 days
Population: All patients with an IVH size greater than 50ml and a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 27 | 28
percentage of participants | 18.5 | 17.9
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.949, Chi-squared; Risk Difference (RD) = 0.0066, 95% CI 2-sided [-0.197 to 0.211]

32. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by Location (Thalamic)
Description: as for outcome 23
Time Frame: 180 days
Population: All patients with a thalamic blood clot location and a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 147 | 139
percentage of participants | 38.8 | 37.4
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.812, Chi-squared; Risk Difference (RD) = 0.014, 95% CI 2-sided [-0.098 to 0.126]

33. Secondary Outcome: Sub-Group Analyses - Difference in Modified Rankin Scale (mRS) 0-3 Proportion by Location (Non-Thalamic)
Description: as for outcome 23
Time Frame: 180 days
Population: All patients with a non-thalamic blood clot location and a non-missing mRS score at 180 days were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 99 | 106
percentage of participants | 60.6 | 54.7
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.394, Chi-squared; Risk Difference (RD) = 0.059, 95% CI 2-sided [-0.076 to 0.194]

34. Secondary Outcome: Functional Status - Barthel Index
Description: Assessment of NIHSS, Barthel Index, eGOS (dichotomy and ordinal) by group. The Barthel Index (BI) assesses ten functional tasks of daily living, and each task provides a measure for level of independence. Scores range from 0 and 100, with a higher score indicating greater independence.
Time Frame: 180 days
Population: All the non-missing Barthel scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: Barthel score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 197 | 170
Barthel score | 65.2 (37.7) | 69.5 (35.1)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.312, Wilcoxon (Mann-Whitney)

35. Secondary Outcome: Functional Status - Participants With Extended Glasgow Outcome (eGOS) Score >=Upper Severe Disability
Description: Assessment of NIHSS, Barthel Index, eGOS (dichotomy and ordinal) by group. The extended Glasgow Outcome Scale (eGOS) is a global scale for functional outcome with eight categories: 1 - Death, 2 - Vegetative State, 3 - Lower Severe Disability, 4 - Upper Severe Disability, 5 - Lower Moderate Disability, 6 - Upper Moderate Disability, 7 - Lower Good Recovery, 8 - Upper Good Recovery.
Time Frame: 180 days
Population: All the non-missing eGOS scores at 180 days were analyzed.
Measure: Number; unit: % of participants with score>=4
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 241 | 241
% of participants with score>=4 | 95 | 77
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.087, Chi-squared — Analysis of dichotomous eGOS, comparing Upper Severe Disability scores to Lower Severe Disability scores; Risk Difference (RD) = 0.075, 95% CI 2-sided [-0.011 to 0.160]
Statistical Analysis 2: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.064, Multivariable Logit Model — Adjusted Multivariable Logit Model comparing eGOS scores of Upper Severe Disability or greater versus Lower Severe Disability and worse; Alteplase versus Saline; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.98 to 2.43]
Statistical Analysis 3: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.336, Generalized Ordered Logit Model — Adjusted generalized ordered logit model odds ratios for eGOS scores of Moderate Disability or worse versus Good Recovery; Alteplase versus Saline; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.70 to 2.89]
Statistical Analysis 4: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.783, Generalized Ordered Logit Model — Adjusted generalized ordered logit model odds ratios for eGOS scores of Upper Severe Disability or worse versus Moderate Disability + Good Recovery; Alteplase versus Saline; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.57 to 1.52]

36. Secondary Outcome: Functional Status - National Institutes of Health Stroke Scale (NIHSS)
Description: Assessment of NIHSS, Barthel Index, eGOS (dichotomy and ordinal) by group. The National Institutes of Health Stroke Scale (NIHSS) is a 15-item scale that assesses language, motor function, sensory loss, consciousness, visual fields, extraocular movements, coordination, neglect, and speech. It is scored from 0 (no stroke symptoms) to 42 (severe stroke).
Time Frame: 180 days
Population: All the non-missing NIHSS scores at 180 days were analyzed.
Measure: Median (Inter-Quartile Range); unit: NIHSS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 182 | 158
NIHSS score | 3 [0 to 9] | 2 [0 to 7]
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.14, Wilcoxon (Mann-Whitney)

37. Secondary Outcome: Quality of Life - Stroke Impact Scale (SIS) - Strength
Description: Assessment of SIS and EuroQol Visual Analog Scale by group. The Stroke Impact Scale (SIS) covers 8 dimensions of stroke outcomes: strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion, memory and thinking, participation. It is scored on a scale of 0 to 100 for each dimension, with higher scores indicating better self-reported health.
Time Frame: 180 days
Population: All the non-missing SIS scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: SIS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 186 | 165
SIS score | 54.97 (35.37) | 58.75 (34.36)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.312, t-test, 2 sided

38. Secondary Outcome: Quality of Life - Stroke Impact Scale (SIS) - Mobility
Description: as for outcome 37
Time Frame: 180 days
Population: All the non-missing SIS scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: SIS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 186 | 165
SIS score | 58.30 (38.16) | 60.10 (36.05)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.65, t-test, 2 sided

39. Secondary Outcome: Quality of Life - Stroke Impact Scale (SIS) - Hand Function
Description: as for outcome 37
Time Frame: 180 days
Population: All the non-missing SIS scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: SIS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 186 | 165
SIS score | 53.41 (41.86) | 56.52 (39.69)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.478, t-test, 2 sided

40. Secondary Outcome: Quality of Life - Stroke Impact Scale (SIS) - Activities of Daily Living
Description: as for outcome 37
Time Frame: 180 days
Population: All the non-missing SIS scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: SIS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 186 | 165
SIS score | 59.33 (37.90) | 61.19 (34.98)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.634, t-test, 2 sided

41. Secondary Outcome: Quality of Life - Stroke Impact Scale (SIS) - Communication
Description: as for outcome 37
Time Frame: 180 days
Population: All the non-missing SIS scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: SIS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 185 | 165
SIS score | 76.02 (31.47) | 79.60 (26.76)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.255, t-test, 2 sided

42. Secondary Outcome: Quality of Life - Stroke Impact Scale (SIS) - Thinking
Description: as for outcome 37
Time Frame: 180 days
Population: All the non-missing SIS scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: SIS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 185 | 165
SIS score | 58.48 (33.11) | 62.68 (31.18)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.224, t-test, 2 sided

43. Secondary Outcome: Quality of Life - Stroke Impact Scale (SIS) - Emotion
Description: as for outcome 37
Time Frame: 180 days
Population: All the non-missing SIS scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: SIS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 185 | 163
SIS score | 73.14 (19.62) | 73.45 (20.24)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.882, t-test, 2 sided

44. Secondary Outcome: Quality of Life - Stroke Impact Scale (SIS) - Participation
Description: as for outcome 37
Time Frame: 180 days
Population: All the non-missing SIS scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: SIS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 186 | 163
SIS score | 47.46 (33.01) | 49.58 (33.03)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.551, t-test, 2 sided

45. Secondary Outcome: Quality of Life - Stroke Impact Scale (SIS) - Recovery
Description: as for outcome 37
Time Frame: 180 days
Population: All the non-missing SIS scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: SIS score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 185 | 162
SIS score | 60.04 (26.42) | 63.44 (25.44)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.224, t-test, 2 sided

46. Secondary Outcome: Quality of Life - EuroQol Visual Analogue Scale (EQ-VAS)
Description: Assessment of SIS and EuroQol Visual Analog Scale by group. EuroQol Visual Analogue Scale (EQ-VAS) is a self-reported measure of health status. It is a marked scale where individuals draw a line to indicate their health, with end points of 0 (the worst health you can imagine) and 100 (the best health you can imagine).
Time Frame: 180 days
Population: All the non-missing EuroQol scores at 180 days were analyzed.
Measure: Mean (Standard Deviation); unit: EuroQol score
Arm/Group | Alteplase | Saline Placebo
Number analyzed (Participants) | 177 | 160
EuroQol score | 62.8 (26.0) | 65.1 (23.3)
Statistical Analysis 1: Comparison: Alteplase vs Saline Placebo; Test type: Superiority or Other; p = 0.376, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 180 days since symptom onset
Arm/Group | Alteplase | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 114/249 | 151/251
Other Adverse Events (participants affected / at risk) | 165/249 | 178/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alteplase (N=249) | Saline Placebo (N=251)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Anoxic brain damage (Nervous system disorders) | 1 (1) | 1 (1)
Anoxic brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Asystole (Cardiac disorders) | 2 (2) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Brain and catheter related infection (Nervous system disorders) | 1 (1) | 0 (0)
Brainstorming/autonomic dysfunction (Nervous system disorders) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 5 (5) | 9 (9)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 3 (3)
Cerebrovascular death (brain death) (Nervous system disorders) | 2 (2) | 6 (6)
Cerebrovascular death (brain death) (General disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Death due to index bleeding event (Nervous system disorders) | 1 (1) | 0 (0)
Death due to index bleeding event (General disorders) | 10 (10) | 21 (21)
Deep vein thrombosis (Vascular disorders) | 6 (6) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 7 (7) | 3 (3)
Depression (Psychiatric disorders) | 1 (3) | 0 (0)
Diabetes mellitus, Type I (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diencephalic storming (Nervous system disorders) | 1 (1) | 0 (0)
Duodenal hemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Edema cerebral (Nervous system disorders) | 3 (3) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Extensor posturing (Nervous system disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Herniation (Nervous system disorders) | 1 (1) | 2 (2)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus, communicating (Nervous system disorders) | 14 (14) | 13 (13)
Hydrocephalus, obstructive (Nervous system disorders) | 1 (1) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
INR increased (Investigations) | 0 (0) | 4 (4)
Intercardiac clot (Cardiac disorders) | 1 (1) | 0 (0)
Interstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Intracranial abcess (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial hemorrhage: Catheter Tract, Enlargement (Nervous system disorders) | 2 (2) | 1 (1)
Intracranial hemorrhage: Catheter Tract, New (Nervous system disorders) | 8 (9) | 7 (7)
Intracranial hemorrhage: Hematoma, subdural (Nervous system disorders) | 1 (2) | 2 (2)
Intracranial hemorrhage: Subarachnoid Space, New (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial hemorrhage: Tissue, Enlargement (Nervous system disorders) | 1 (1) | 1 (1)
Intracranial hemorrhage: Tissue, New (Nervous system disorders) | 2 (2) | 5 (5)
Intracranial hemorrhage: Ventricular system, Enlargement (Nervous system disorders) | 3 (3) | 2 (2)
Intracranial hemorrhage: Ventricular system, New (Nervous system disorders) | 2 (2) | 3 (3)
Intracranial hypertension (Nervous system disorders) | 9 (9) | 8 (11)
Intrahepatic cholestasis of unk etiology (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 3 (3) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Meningitis (Nervous system disorders) | 2 (2) | 3 (3)
Multi-organ failure (General disorders) | 1 (1) | 3 (3)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
PEG Tube complication (Surgical and medical procedures) | 1 (1) | 0 (0)
Peritoneal infection (Infections and infestations) | 0 (0) | 2 (2)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 13 (14)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal insufficiency (Renal and urinary disorders) | 6 (6) | 6 (6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 17 (17)
Reversible cerebral vasoconstriction vs vasculitis (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 11 (13) | 7 (8)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Stroke (Nervous system disorders) | 4 (4) | 4 (4)
Sudden death NOS (General disorders) | 6 (6) | 8 (8)
Supraventricular tachydysrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Takotsubo syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 8 (9)
VP shunt dysfunction (Nervous system disorders) | 1 (1) | 1 (1)
Vasospasm or DIND (Nervous system disorders) | 2 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Ventriculitis, bacterial (Infections and infestations) | 1 (1) | 1 (1)
Ventriculitis, bacterial (Nervous system disorders) | 3 (3) | 10 (12)
Ventriculitis, non-bacterial (Infections and infestations) | 1 (1) | 0 (0)
Ventriculitis, non-bacterial (Nervous system disorders) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound infection, non-neurologic (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alteplase (N=249) | Saline Placebo (N=251)
Bacteremia (Infections and infestations) | 13 (13) | 6 (7)
Deep vein thrombosis (Vascular disorders) | 21 (21) | 20 (20)
Depressed level of consciousness (Nervous system disorders) | 6 (7) | 12 (13)
Fever (General disorders) | 72 (76) | 67 (74)
Hydrocephalus, communicating (Nervous system disorders) | 24 (24) | 33 (33)
Intracranial hemorrhage: Catheter Tract, New (Nervous system disorders) | 34 (37) | 39 (47)
Intracranial hypertension (Nervous system disorders) | 39 (53) | 42 (50)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 41 (41) | 53 (53)
Seizure (Nervous system disorders) | 13 (14) | 16 (20)
Urinary tract infection (Infections and infestations) | 36 (38) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes